CLINICAL TRIAL: NCT04816279
Title: Clinical Audit on the Quality of Care of Elective Caesarean Section
Brief Title: Enhanced Recovery After Cesarean Section
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Youstina Tharwat Adeeb, Dr, Assiut University
Other Study IDs: CAQOCACS
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Cesarean Section; Quality Of Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First Audit cycle
- Second Audit cycle

SUMMARY:
1. Measure compliance of the care of elective caesarean section with ERAS standards
2. Measure the quality of recovery of women undergoing elective caesarean section

DETAILED DESCRIPTION:
Caesarean section is one of most common surgeries worldwide and in Egypt. The Egyptian Demographic and Health Survey 2014 revealed a rising caesarean section rate .

Many of these procedures are elective allowing time for preparation of the patient for surgery.

Enhanced recovery after surgery (ERAS) is a multimodal, multi disciplinary, evidence based approach to surgical care with an ultimate goal to enhance recovery and improve maternal and neonatal outcome .

This is done through optimizing multiple aspects of patient care to enhance recovery and so accelerate (facilitate) earlier discharge (decrease length of stay, decrease opioids use and encourage breastfeeding) .

A comparative study in Egypt found ERAS to be effective in controlling perioperative gastrointestinal symptoms, pain control and encourages early ambulation with offering earlier resumption of intestinal motility, higher satisfaction and fewer days of admission .

The clinical audit is a tool for assessing the compliance of current practice with the standard of care. In an audit, both process of care compliance and outcome of care can be measured to highlight gaps that need to be addressed by the institution . Enhanced Recovery After Surgery society issued Guidelines for elective Cesarean Section care .

They include elements in preoperative, intraoperative and postoperative care. Compliance with each of these items was associated with improved maternal or neonatal outcome and a better recovery experience .

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing elective caesarean section in the study period

Exclusion Criteria:

* Women who cannot apply ERAS protocol

  1. emergency caesarean section
  2. anticipated surgical difficulty e.g. placenta previa/accrete, tumors obstructing lower uterine segment
  3. Severe maternal disease
  4. severe intraoperative bleeding or visceral injuries necessitating modification of postoperative care

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: women undergoing scheduled and arranged cesarean sections
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
the percentage of compliance of care with ERAS society guidelines | baseline
  compliance of routinely provided care with ERAS society guidelines

SECONDARY OUTCOMES:
Quality of recovery after elective caesarean section | baseline
  better recovery experience with less length of stay at hospital

REFERENCES:
- [Background] Kleiman AM, Chisholm CA, Dixon AJ, Sariosek BM, Thiele RH, Hedrick TL, Carvalho B, Tiouririne M. Evaluation of the impact of enhanced recovery after surgery protocol implementation on maternal outcomes following elective cesarean delivery. Int J Obstet Anesth. 2020 Aug;43:39-46. doi: 10.1016/j.ijoa.2019.08.004. Epub 2019 Aug 21. PMID 31522935
- [Background] Mullman L, Hilden P, Goral J, Gwacham N, Tauro C, Spinola K, Rosales K, Collier S, Holmes L, Maccione J, Pitera R, Miller R, Yodice P. Improved Outcomes With an Enhanced Recovery Approach to Cesarean Delivery. Obstet Gynecol. 2020 Oct;136(4):685-691. doi: 10.1097/AOG.0000000000004023. PMID 32925620
- [Background] Tan HS, Habib AS. The optimum management of nausea and vomiting during and after cesarean delivery. Best Pract Res Clin Anaesthesiol. 2020 Dec;34(4):735-747. doi: 10.1016/j.bpa.2020.04.012. Epub 2020 Apr 23. PMID 33288123
- [Background] Wilson RD, Caughey AB, Wood SL, Macones GA, Wrench IJ, Huang J, Norman M, Pettersson K, Fawcett WJ, Shalabi MM, Metcalfe A, Gramlich L, Nelson G. Guidelines for Antenatal and Preoperative care in Cesarean Delivery: Enhanced Recovery After Surgery Society Recommendations (Part 1). Am J Obstet Gynecol. 2018 Dec;219(6):523.e1-523.e15. doi: 10.1016/j.ajog.2018.09.015. Epub 2018 Sep 18. PMID 30240657
- [Background] Caughey AB, Wood SL, Macones GA, Wrench IJ, Huang J, Norman M, Pettersson K, Fawcett WJ, Shalabi MM, Metcalfe A, Gramlich L, Nelson G, Wilson RD. Guidelines for intraoperative care in cesarean delivery: Enhanced Recovery After Surgery Society Recommendations (Part 2). Am J Obstet Gynecol. 2018 Dec;219(6):533-544. doi: 10.1016/j.ajog.2018.08.006. Epub 2018 Aug 15. PMID 30118692
- [Background] Macones GA, Caughey AB, Wood SL, Wrench IJ, Huang J, Norman M, Pettersson K, Fawcett WJ, Shalabi MM, Metcalfe A, Gramlich L, Nelson G, Wilson RD. Guidelines for postoperative care in cesarean delivery: Enhanced Recovery After Surgery (ERAS) Society recommendations (part 3). Am J Obstet Gynecol. 2019 Sep;221(3):247.e1-247.e9. doi: 10.1016/j.ajog.2019.04.012. Epub 2019 Apr 14. PMID 30995461
- [Background] From the American Association of Neurological Surgeons (AANS), American Society of Neuroradiology (ASNR), Cardiovascular and Interventional Radiology Society of Europe (CIRSE), Canadian Interventional Radiology Association (CIRA), Congress of Neurological Surgeons (CNS), European Society of Minimally Invasive Neurological Therapy (ESMINT), European Society of Neuroradiology (ESNR), European Stroke Organization (ESO), Society for Cardiovascular Angiography and Interventions (SCAI), Society of Interventional Radiology (SIR), Society of NeuroInterventional Surgery (SNIS), and World Stroke Organization (WSO); Sacks D, Baxter B, Campbell BCV, Carpenter JS, Cognard C, Dippel D, Eesa M, Fischer U, Hausegger K, Hirsch JA, Shazam Hussain M, Jansen O, Jayaraman MV, Khalessi AA, Kluck BW, Lavine S, Meyers PM, Ramee S, Rufenacht DA, Schirmer CM, Vorwerk D. Multisociety Consensus Quality Improvement Revised Consensus Statement for Endovascular Therapy of Acute Ischemic Stroke. Int J Stroke. 2018 Aug;13(6):612-632. doi: 10.1177/1747493018778713. Epub 2018 May 22. No abstract available. PMID 29786478